CLINICAL TRIAL: NCT03783598
Title: Person-Centered, Occupation Based Intervention Program Supported With Problem-Solving Therapy for Type 2 Diabetes
Brief Title: Person-Centered, Occupation Based Therapy for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, ZEYNEP BAHADIR AGCE, Assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 569831°
Record Dates: First submitted 2018-12-14; First posted 2018-12-21 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2; Occupational Therapy
Keywords: Diabetes Mellitus; Problem Solving; Occupational Therapy; Healthy Lifestyle; Occupational Performance; Person-Centered; Occupation Based
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: The problem solving therapy is an social cognitive therapy approach. And ıt support to solve meaningfull occupational performance problems realted to diabetes by invdividuals and this way, it helps to improve the self-management of diabetes.We used that with person centered perspective and support to person with education which was perspective of person environment occupation model.
Who Masked: Participant
Masking Description: The study population was 76 individuals whose diagnosis of type 2 diabetes. 9 volunteer individual gave up to participation without for various reasons in the process.That intervention grup (n=33) control group (n=34), between the ages of 18 to 65 years and volunteer individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group received problem solving therapy as 6 modules. Each module was included at least 1 session per week that is nearly 60 minutes, and the amount of weekly sessions was arranged according to the needs of the person.Individuals has an opportunity was provided for identify problems meaningful for themselves and to start their change from the activities they valued by using the COPM.
  Interventions: Behavioral: Person centered, occupation based intervention support with problem solving therapy
- control group (No Intervention): Control group had not any intervention we have an education to control group about diabetes and healthy life conditions.

INTERVENTIONS:
Behavioral: Person centered, occupation based intervention support with problem solving therapy — This program that was developed from the occupational therapy perspective which is person centered and occupation based for T2D intervention was designed as 6 modules. The intervention group received person centered, occupation based intervention support with problem solving therapy as 6 modules. The control group had not any intervention, just had a education about effect of diabetes on life.
  Other Names: self management
  Arms: intervention group

SUMMARY:
This study was conducted to investigate the effect of a person-centered, occupation-based intervention program supported with problem-solving strategy in individuals with type 2 diabetes (T2D).

Method: The study was a randomized controlled trial, that included intervention (n=33) and control group (n=34), between the ages of 18 and 65 years.

DETAILED DESCRIPTION:
It was planned as a single-blind, randomized controlled study with 3-month follow-up in adults. A total of 67 subjects were randomly allocated to the intervention (n=33) or the control group (n=34). This program prepared with consider to meaningful activities for individual and overcome to barriers via problem solving. That was designed as 6 modules including evaluations, diabetes education and problem-solving therapy. Each module was implemented at least 1 session per week, about 60 minutes, and was arranged according to individual needs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Able to read and write turkish

Exclusion Criteria:

* Cancer
* Mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Canada activity performance measure (COPM) | Intervention and control groups' each participants were analyze before the intervention modules with assessment tools. All assessment tools repeated 6 weeks and 3 months later from the intervention modules.
  COPM, measure self-perceived change in problem on occupational performance and satisfaction over time. The COPM enable individuals to identify and prioritize everyday issues that restrict or impact their performance in everyday living. In the first step, occupational therapist interviews with client determine what the individual has done in his/her routine, what he/she wants to do or can not to do in their self-care, productivity and free time. Secondly the client to rate, on a scale of 1 to 10, the importance of each activity. Then confirming with the client the 5 most important problems and record. The client to rate each problem on performance and satisfaction, then calculate the total scores.
  Total scores are calculated by adding together the performance or satisfaction scores for all problems and dividing by the number of problems. At reassessment,the client scores each problem again for performance and satisfaction. Calculate the new scores and the change score.

SECONDARY OUTCOMES:
The diabetes empowerment scale (DES) | Intervention and control groups' each participants were analyze before the intervention modules with assessment tools. All assessment tools repeated 6 weeks and 3 months later from the intervention modules.
  DES measure the psychosocial self-efficacy of people with diabetes. The scale consists of three factors; managing the psychosocial aspects of diabetes (9 items), assessing dissatisfaction and readiness to change (9 items), setting and achieving diabetes goals (10 items). Each question on the diabetes empowerment scale scores between 1 (strongly disagree) to 5 (strongly agree). The total score of the scale, calculated by adding all of the item scores and dividing by 28. High score indicates that the levels of empowerment are high.
The Brief COPE | Intervention and control groups' each participants were analyze before the intervention modules with assessment tools. All assessment tools repeated 6 weeks and 3 months later from the intervention modules.
  The Brief COPE assess coping style with stress. Brief COPE include 14 subscale such as self-distraction (items 1 and 19), active coping, (items 2 and 7), denial, (items 3 and 8), substance use, (items 4 and 11), use of emotional support, (items 5 and 15), use of instrumental support, (items 10 and 23), behavioral disengagement, (items 6 and 16),venting, (items 9 and 21), positive reframing, items 12 and 17), planning, (items 14 and 25),humor, (items 18 and 28). each options rate range from 1 (ı'm not doing this at all) to 4 (ı'm doing this a lot), and min-max score range from 2 to 8.
WHO-five well-being index (WHO-5) | Intervention and control groups' each participants were analyze before the intervention modules with assessment tools. All assessment tools repeated 6 weeks and 3 months later from the intervention modules.
  The WHO-5 well being index was used to psychometrically sound measure of emotional well-being. The answer for each question are given considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The total score changes to ranges from 0 (absence of well-being) to 25 (maximum well-being). The raw score is multiplied by 4 to obtain a percentage score between 0 and 100. When the changes is 10% in raw score, that indicates a significant change.
Demographic questionnaire | Before the intervention
  Demographic questionnaire: At first all participants filled a questionnaire covering demographic form, which included the participant's age, gender, education, health habits (smoking, alcohol consumption, participation in sport) and body mass index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP B BAHADIR AGCE, PHD, Study Director — occupational therapy
Locations (2):
- Turkey (Türkiye) (2):
  - Gamze Ekici Çağlar, Ankara
  - Zeynep Bahadır Ağce, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weigensberg MJ, Vigen C, Sequeira P, Spruijt-Metz D, Juarez M, Florindez D, Provisor J, Peters A, Pyatak EA. Diabetes Empowerment Council: Integrative Pilot Intervention for Transitioning Young Adults With Type 1 Diabetes. Glob Adv Health Med. 2018 Mar 8;7:2164956118761808. doi: 10.1177/2164956118761808. eCollection 2018. PMID 29552422
- [Background] Hill-Briggs F. Problem solving in diabetes self-management: a model of chronic illness self-management behavior. Ann Behav Med. 2003 Summer;25(3):182-93. doi: 10.1207/S15324796ABM2503_04. PMID 12763713
- [Result] Hwang JE, Truax C, Claire M, Caytap AL. Occupational therapy in diabetic care-areas of need perceived by older adults with diabetes. Occup Ther Health Care. 2009;23(3):173-88. doi: 10.1080/07380570902950259. PMID 23927025
- [Derived] Bahadir Agce Z, Ekici G. Person-centred, occupation-based intervention program supported with problem-solving therapy for type 2 diabetes: a randomized controlled trial. Health Qual Life Outcomes. 2020 Aug 3;18(1):265. doi: 10.1186/s12955-020-01521-x. PMID 32746841